CLINICAL TRIAL: NCT04472897
Title: A Randomised, Double Blind (Sponsor Unblinded), Placebo-controlled, First Time in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Oral Doses and the Food Effect of GSK2556286 in Healthy Adult Participants
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of GSK2556286 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A decision to stop the study was made by the site and GSK project team based on pre-defined stopping criteria in the protocol
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 210035
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis
Keywords: GSK2556286; Pharmacokinetics; Interventional; Tuberculosis; Placebo-controlled; First time in human
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, sequential, parallel dose cohort study.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Participants receiving GSK2556286 (Experimental): Participants will be randomized to receive GSK2556286 in any of the 11 cohorts. In each dosing cohort, 6 participants will receive a single dose of GSK2556286. Following initial dosing of cohorts in the fasted state, one cohort will investigate the effect of food administration (high fat meal) on safety, tolerability and PK data of GSK2556286. One cohort may also investigate the effects of a moderate fat meal.
  Interventions: Drug: GSK2556286
- Part A: Participants receiving placebo (Placebo Comparator): Participants will be randomized to receive matching placebo in any of the 11 cohorts. In each dosing cohort, 2 participants will receive a single dose of matching placebo.
  Interventions: Drug: Placebo
- Part B: Participants receiving GSK2556286 (Experimental): Participants will be randomized to receive GSK2556286 in any of the 4 cohorts. In each dosing cohort, 6 participants will receive repeat doses of GSK2556286 under either fasting or fed conditions, dependent on the results from Part A.
  Appropriate doses and dose regimens for Part B will be selected by the Dose Escalation Committee based on available safety, tolerability and PK data from Part A and/or any preceding repeat dose cohorts from Part B.
  Interventions: Drug: GSK2556286
- Part B: Participants receiving placebo (Placebo Comparator): Participants will be randomized to receive matching placebo in any of the 4 cohorts. In each dosing cohort, 2 participants will receive repeat doses of matching placebo under either fasting or fed conditions, dependent on the results from Part A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2556286 — GSK2556286 will be administered.
  Arms: Part A: Participants receiving GSK2556286; Part B: Participants receiving GSK2556286
Drug: Placebo — Placebo will be administered
  Arms: Part A: Participants receiving placebo; Part B: Participants receiving placebo

SUMMARY:
This first time in human (FTIH) study assesses the safety, tolerability, and pharmacokinetics (PK) of single and multiple increasing doses of GSK2556286. It also includes food effect cohorts to evaluate how food influences the PK of GSK2556286. The findings will help determine appropriate dosing for future clinical studies.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 60 years of age inclusive, at the time of signing the informed consent. Participants aged 51 to 60 years must have received at least one dose of Coronavirus disease-2019 (COVID-19) vaccine approved by the local regulatory authority at least 3 weeks prior to signing the consent form.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included only if the Investigator considers and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight more than or equal to (>=)50 kilograms (kg) and body mass index (BMI) within the range 19 to 29.9 kilograms per meter square (kg/m^2) inclusive.
* Male and/or Female Participants. A male participant with a female partner of reproductive potential must agree to use contraception of this clinical study protocol during the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period. A female participant is eligible to participate if she is not a woman of childbearing potential (WONCBP).
* The participant is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion criteria:

* Significant history of or current, cardiovascular, respiratory (including asthma), hepatic, renal, gastrointestinal, endocrine, hematological, infectious or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs: constituting a risk when taking part in the study or interfering with the interpretation of data.
* Alanine aminotransferase (ALT) greater than (>)1.5 times upper limit of normal (ULN).
* Total bilirubin >1.5 times ULN (isolated total bilirubin >1.5 times ULN may be acceptable, after consultation with the GlaxoSmithKline (GSK) Medical Monitor, if total bilirubin is fractionated and direct bilirubin less than [<]35 percent [%]).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or cholecystectomy.
* Current or past history of significant renal disease including renal stones.
* Current or past history of gastroduodenal ulcers or persistent gastritis requiring medication.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Exclusion criteria for screening electrocardiogram (ECG) with:

  1. Heart rate of <40 or >100 beats per minute (bpm) in males and <50 or >100 bpm in females.
  2. PR interval of <120 or >220 milliseconds (msec) in males and females.
  3. QRS duration of <70 or >120 msec in males and females.
  4. Electrocardiogram QT interval corrected for heart rate using Fridericia's formula (QTcF) interval of >450 msec in males and females.
* Evidence of previous myocardial infarction (does not include ST segment changes associated with re-polarization).
* Any clinically significant conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular [AV] block [second degree or higher], Wolff -Parkinson-White [WPW] syndrome).
* Sinus Pauses >3 seconds.
* Any significant arrhythmia which, in the opinion of the Investigator or GSK Medical monitor, will interfere with the safety for the individual participant.
* Non-sustained or sustained ventricular tachycardia (3 consecutive ventricular ectopic beats).
* Evidence of latent tuberculosis documented by:

  1. medical history and examination.
  2. Tuberculosis (TB) testing : either a positive tuberculin skin test (TST) (defined as a skin induration >5 millimeters [mm] at 48 to 72 hours, regardless of Bacillus Calmette-Guerin (BCG) or other vaccination history) or a positive (not indeterminate) TB test such as QuantiFERON-TB Gold Plus test. In cases where the QuantiFERON or TST is indeterminate, the participant may have the test repeated once, but they will not be eligible for the study unless the second test is negative. In cases where the QuantiFERON or TST test is positive, the participant should be followed up as per standard of care.
* Use of prescription or non-prescription drugs, including Nonsteroidal anti-inflammatory drugs (NSAIDs), high-dose vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Cotinine in urine indicative of smoking or history or regular use of tobacco or nicotine-containing products within 3 months.
* Current regular alcohol consumption defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive test for Human immunodeficiency virus (HIV) antibody.
* Urinary analysis indicating presence of blood, protein or glucose. If trace or 1 plus (+) is found on urine dipstick, a repeat test can be performed. If repeat is positive, participant is excluded from recruitment.
* Screening age-appropriate estimated glomerular filtration rate (eGFR) <90 milliliters per minute mL/min as assessed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Serum (and in the MAD, urinary) electrolytes outside of normal range. May be repeated once if abnormal.
* A positive pre-study drug/alcohol screen.
* The participant has taken part in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Part A (Food Effect) Cohort: Participant must have no relevant dietary restrictions (lactose intolerance) or inability to eat a high fat meal.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with any serious adverse events (SAEs) and non-SAEs | Up to Day 15
Part B: Number of participants with any SAEs and non-SAEs | Up to Day 28
Part A: Number of participants with AEs (SAEs and non-SAEs) by severity | Up to Day 15
Part B: Number of participants with AEs (SAEs and non-SAEs) by severity | Up to Day 28
Part A: Plasma concentrations of GSK2556286 | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Area under the plasma drug concentration versus time curve from time zero to last time of quantifiable concentration (AUC[0-t]) of GSK2556286 | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: AUC from time zero extrapolated to infinity (AUC[0-inf]) of GSK2556286 | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Maximum observed plasma drug concentration (Cmax) of GSK2556286 | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Time to maximum observed plasma drug concentration (Tmax) of GSK2556286 | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Apparent terminal half-life (T1/2) of GSK2556286 | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Plasma concentrations of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose. Day 12 and 13: Pre-dose
Part B: AUC(0-t) of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: AUC(0-inf) of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Area under the plasma drug concentration versus time curve from time zero during a dosage interval of time tau (AUC[0-tau)] of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Cmax of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Tmax of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Trough plasma concentration (Ctau) of GSK2556286 | Pre-dose on Days 1, 12, 13 and 14
Part B: T1/2 of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose

SECONDARY OUTCOMES:
Part A: AUC(0-t) of GSK2556286 under fasted and fed conditions | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: AUC(0-inf) of GSK2556286 under fasted and fed conditions | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Cmax of GSK2556286 under fasted and fed conditions | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Tmax of GSK2556286 under fasted and fed conditions | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: T1/2 of GSK2556286 under fasted and fed conditions | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Dose proportionality of GSK2556286 based on AUC(0-inf) | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Dose proportionality of GSK2556286 based on AUC(0-t) | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part A: Dose proportionality of GSK2556286 based on Cmax | Day 1: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Dose proportionality of GSK2556286 based on AUC(0-tau) | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Dose proportionality of GSK2556286 based on Cmax | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Observed accumulation ratio of GSK2556286 based on AUC (AUC[Ro]) | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Observed accumulation ratio of GSK2556286 based on Cmax (RCmax) | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Steady state ratio (Rss) of GSK2556286 | Day 1 and 14: Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48 and 72 hours post-dose
Part B: Ctau at the end of the dosing interval to assess steady state of GSK2556286 | Pre-dose on Days 1, 12, 13 and 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Groningen, Netherlands
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Nuermberger EL, Martinez-Martinez MS, Sanz O, Urones B, Esquivias J, Soni H, Tasneen R, Tyagi S, Li SY, Converse PJ, Boshoff HI, Robertson GT, Besra GS, Abrahams KA, Upton AM, Mdluli K, Boyle GW, Turner S, Fotouhi N, Cammack NC, Siles JM, Alonso M, Escribano J, Lelievre J, Rullas-Trincado J, Perez-Herran E, Bates RH, Maher-Edwards G, Barros D, Ballell L, Jimenez E. GSK2556286 Is a Novel Antitubercular Drug Candidate Effective In Vivo with the Potential To Shorten Tuberculosis Treatment. Antimicrob Agents Chemother. 2022 Jun 21;66(6):e0013222. doi: 10.1128/aac.00132-22. Epub 2022 May 24. PMID 35607978